CLINICAL TRIAL: NCT03917316
Title: Language and Narrative Abilities of Children With ADHD and the Association to Executive Function, ADHD Symptoms and Social and Academic Function
Brief Title: Language Abilities of Children With ADHD
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Language and ADHD
Record Dates: First submitted 2019-04-04; First posted 2019-04-17 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ADHD
  Interventions: Other: Language and neuropsychological tests
- Control
  Interventions: Other: Language and neuropsychological tests

INTERVENTIONS:
Other: Language and neuropsychological tests — Tests related to language, narrative and specific and general cognitive function

SUMMARY:
BACKGROUND: Attention-Deficit/Hyperactivity-Disorder (ADHD) is associated with language difficulties within expressive, receptive and pragmatic areas of language.Telling stories is a particularly interesting language task as is provides the possibility of investigating how children use their language in everyday interactions. Thus, investigating how children with ADHD tell stories provides a more naturalistic impression of their language abilities. However, the extent, causes, and clinical relevance of language and narrative difficulties in ADHD remain largely unknown. Language may be the key to understanding and improving the functional impairments associated with ADHD such as social and academic function.

AIM: The overall aim of the current study was to investigate the association between language, narrative ability and ADHD, what contributes to this association, as well as the clinical relevance of language difficulties in ADHD in relation to academic and social function.

METHOD: Children between 7-11 years old with ADHD will be recruited from Aarhus University Hospital in Skejby and compared to children without ADHD recruited from schools in the community. All children will be assessed at two separate meetings at the Department of Psychology, Aarhus University. The total number of participants in each group will depend on the intake of patients at Aarhus University Hospital, but a maximum of 100 children will be sampled in each group.

DETAILED DESCRIPTION:
BACKGROUND:

Up to 40% of children with the ADHD are suggested to have language difficulties. Other than language difficulties being debilitating in their own right, language difficulties in childhood ADHD are problematic because they likely enhance the social and academic difficulties often present in children with this disorder. Children with ADHD also appear to have narrative difficulties; i.e. they have problems telling a coherent, understandable story. Telling stories is a particularly interesting language task as the investigation of how children use their language in an unstructured task is similar to how they use their language in everyday interactions.

However, the extent, causes, and clinical relevance of language and narrative difficulties in ADHD remain largely unknown. Studies are scarce and fraught with problems warranting investigations of language abilities in children with ADHD that measure language as well as executive function (EF) and that investigate the clinical relevance of these language difficulties. This is necessary in order to tease apart and gain knowledge of the association between language, EF and ADHD. Ultimately, such an investigation can inspire future assessment and treatment of language difficulties in children with ADHD.

AIMS AND HYPOTHESES

1. The first aim is to examine narrative abilities in children with ADHD. This is done by investigating whether children with and without ADHD differ with respect to their narratives.
2. The second aim is to examine whether language, EF and/or ADHD symptoms can explain narrative function in children with and without ADHD.
3. The third aim is to investigate which specific domains of language children with ADHD have the most difficulty within.
4. The fourth aim is to investigate whether the language difficulties as well as the narrative difficulties identified are associated with academic and social function in ADHD.

PARTICIPANTS AND PROCEDURES Up to 100 children with ADHD, age 7-11, consecutively referred from Aarhus University Hospital, Denmark, will be compared to up to 100 typically developing children, age 7-11, recruited from schools in the same community as the hospital.

After initial screening by telephone, informed consent has been obtained from both custodians and verbal assent has been given by the child, all children (ADHD and control) will be assessed at two separate meetings at the University of Aarhus by a member of the project group. The parents will receive questionnaires about their child and if the families give their consent, questionnaires will also be sent to the children's primary teacher. The parents and teachers receive questionnaires about the child's behavior, language and social and academic abilities.

All hypotheses will be investigated with appropriate statistical analyses. The role of IQ, parental educational level etc. is also examined in the analyses. If an adequate sample size is obtained, confirmatory factor analysis (CFA) will be applied to handle data, and if a factor solution is supported, factor scores will be included in all analyses, thereby reducing the number of variables in the analyses.

REGISTRATION DETAILS The study record reported at clinical trials.gov is completely consistent with the protocol approved by the Central Region Committee on Health Research Ethics in Denmark. The study was registered at clinical trials.gov after enrollment had begun, but no changes have been made in any procedures, recruitment etc., and as such it was assessed to be feasible to include the few participants that had been enrolled before registration in clinical trials.

ELIGIBILITY:
Inclusion criteria

* Age between 7 and 11 years.
* For the clinical group: Current ADHD diagnosis (Development and Well-Being Assessment; DAWBA, Goodman et al., 2000).

Exclusion criteria:

* Autism spectrum diagnosis (ASD) based on the Development and Well-Being Assessment (DAWBA, Goodman et al., 2000) or a history of ASD based on parent report on a background questionnaire.
* Epilepsy or known brain damage based on parent report (background questionnaire).
* IQ < 70 based on an intelligence test.
* Danish as a second language, based on parent report (background questionnaire).
* Low birth weight (<1500 grams) based on parent report (background questionnaire).
* Premature birth (before 32nd gestation week) based on parent report (background questionnaire).
* Use of medication that is expected to affect cognition (background questionnaire).
* Impaired sight, hearing, or motor function (as this would interfere with task performance), based on parent report (background questionnaire).
* For the control group: Current (based on the DAWBA) or previous (based on parent- reports from the background questionnaire) ADHD diagnosis.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The clinical group of children with ADHD will be recruited from the Aarhus University Hospital and the typical developing control group will be recruited from schools in the community.
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
General language ability | One day
  Clinical Evaluation of Language Fundamentals-4 (Semel, Wiig & Secord, 2003), measures general language ability. Rawscores on the task are converted to scale scores with a range of 1-14. A scale score of 7-10 is average, above indicates better language proficiency.
Pragmatic language ability | One day
  Children's Communication Checklist-2 (CCC-2; Bishop, 2002), index for pragmatic ability, scaled scores (0-14), where 7-10 is average and above indicates better pragmatic language ability.
Narrative abilities | One day
  Online story-telling of the wordless picture book "Frog, where are you"
Working memory 2back task | One day
  A self-designed 2back task modelled from Friedman et al., 2008). Measures the child's working memory. Outcome is mean accuracy, range 0-1, with higher scores indicating better working memory.
Working memory Mental Counters task | One day
  Mental Counters (Huizinga et al., 2006). Measures the child's working memory. Outcome is mean accuracy, range 0-1, with higher scores indicating better working memory.
Working memory Tic Tac Toe task | One day
  Tic Tac Toe (Huizinga et al., 2006). Measures the child's working memory. Outcome is mean accuracy, range 0-1, with higher scores indicating better working memory.
Inhibition Stop-signal task | One day
  Stop-Signal task (Logan 1994; Logan, Schachar & Tannock, 1997; Williams, Pronesse, Schachar; Logan & Tannock, 1999); outcome Stop-signal Reaction time (SSRT), with slower reaction times indicating problems with inhibtion.
Inhibition Flanker task | One day
  Flanker task (Huyser et al., 2011), outcome median reaction time on conflict trials, with higher median reaction times indicating problems within inhibition.
Inhibition Go/No Go task | One day
  Go/No go (Tsujimoto, 2006), outcome percent false alarms, higher percents indicating problems within inhibition.
Social abilities | One day
  Social Competence Inventory-2 (Rydell Hagekull & Bohlin, 1997) a questionnaire about social competencies. The parents rate their child on a scale of 1-5 on 25 questions, higher scores indicate better social ability.
Academic abilities | One day
  5-15 questionnaire (Kadesjö, Janols, Korkman, Mickelsson, Strand, Trillingsgaard & Gillberg, 2005). Questions from the learning domain. The parent rates the child on a scale of 1-3 on 29 questions about academic ability, with higher scores indicating academic difficulties.
Academic abilities teacher | One day
  Teacher Telephone Interview (TTI, Tannock, Manassis & Fung, 2003, revised and translated with permission from R. Tannock). The teacher rates the child on a scale of 1-5 on 9 school subjects. Higher scores indicate better academic ability.
Executive functions | One day
  Childhood Executive Functioning inventory (CHEXI; Nyberg & Thorell, 2008). Questionnaire. The parent rates the child on a scale of 1-5 on 26 questions concerning the childs executive functioning. Higher scores indicate problems within executive functioning.

SECONDARY OUTCOMES:
Reaction time | One day
  Reaction time task (Tsujimoto, 2006) measures the child's average reaction time, with higher scores indicating faster reaction time.
General cognitive abilities | One day
  Ravens Coloured Matrices (Raven, 1998). A task that measures the child's general cognitive ability on a scale of 0-36, where higher scores indicate better cognitive abilities.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, Aarhus University, Aarhus, (non-US), Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellani M, Moretti A, Perlini C, Brambilla P. Language disturbances in ADHD. Epidemiol Psychiatr Sci. 2011 Dec;20(4):311-5. doi: 10.1017/s2045796011000527. PMID 22201208
- [Background] Flory K, Milich R, Lorch EP, Hayden AN, Strange C, Welsh R. Online story comprehension among children with ADHD: which core deficits are involved? J Abnorm Child Psychol. 2006 Dec;34(6):853-65. doi: 10.1007/s10802-006-9070-7. Epub 2006 Oct 19. PMID 17051434
- [Background] Jensen, K. d. L. (2011). Specifik sprogforstyrrelse - en komorbid forstyrrelse ved ADHD Best Practice, 14, 36-37.
- [Background] Korrel H, Mueller KL, Silk T, Anderson V, Sciberras E. Research Review: Language problems in children with Attention-Deficit Hyperactivity Disorder - a systematic meta-analytic review. J Child Psychol Psychiatry. 2017 Jun;58(6):640-654. doi: 10.1111/jcpp.12688. Epub 2017 Feb 10. PMID 28186338
- [Background] Sciberras E, Mueller KL, Efron D, Bisset M, Anderson V, Schilpzand EJ, Jongeling B, Nicholson JM. Language problems in children with ADHD: a community-based study. Pediatrics. 2014 May;133(5):793-800. doi: 10.1542/peds.2013-3355. PMID 24753530
- [Background] Gremillion ML, Martel MM. Semantic language as a mechanism explaining the association between ADHD symptoms and reading and mathematics underachievement. J Abnorm Child Psychol. 2012 Nov;40(8):1339-49. doi: 10.1007/s10802-012-9650-7. PMID 22661106
- [Background] Lambek R, Tannock R, Dalsgaard S, Trillingsgaard A, Damm D, Thomsen PH. Executive dysfunction in school-age children with ADHD. J Atten Disord. 2011 Nov;15(8):646-55. doi: 10.1177/1087054710370935. Epub 2010 Sep 21. PMID 20858784
- [Background] Purvis KL, Tannock R. Language abilities in children with attention deficit hyperactivity disorder, reading disabilities, and normal controls. J Abnorm Child Psychol. 1997 Apr;25(2):133-44. doi: 10.1023/a:1025731529006. PMID 9109030
- [Background] Staikova E, Gomes H, Tartter V, McCabe A, Halperin JM. Pragmatic deficits and social impairment in children with ADHD. J Child Psychol Psychiatry. 2013 Dec;54(12):1275-83. doi: 10.1111/jcpp.12082. Epub 2013 May 18. PMID 23682627
- [Background] Whitely C, Colozzo P. Who's Who? Memory updating and character reference in children's narratives. J Speech Lang Hear Res. 2013 Oct;56(5):1625-36. doi: 10.1044/1092-4388(2013/12-0176). Epub 2013 Jun 19. PMID 23785191